CLINICAL TRIAL: NCT02175199
Title: A Comparison of Two Color Contact Lenses in Habitual Clear Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: M-14-008
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-09

CONDITIONS: Myopia
Keywords: Contact lens; Vision care; Daily wear; Color contact lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR OPTIX COLORS (Experimental): Lotrafilcon B contact lenses with color printing worn bilaterally in a daily wear modality 5 days/week, 8 hours/day for 30 days.
  Interventions: Device: Lotrafilcon B contact lenses with color printing
- FreshLook COLORBLENDS (Active Comparator): Phemfilcon A contact lenses with color printing worn bilaterally in a daily wear modality 5 days/week, 8 hours/day for 30 days with a 2-week replacement.
  Interventions: Device: Phemfilcon A contact lenses with color printing

INTERVENTIONS:
Device: Lotrafilcon B contact lenses with color printing
  Other Names: AIR OPTIX® COLORS
  Arms: AIR OPTIX COLORS
Device: Phemfilcon A contact lenses with color printing
  Other Names: FreshLook® COLORBLENDS®
  Arms: FreshLook COLORBLENDS

SUMMARY:
The purpose of this study is to evaluate the comfort of color contact lenses in a population of clear contact lens wearers who have an interest in wearing color contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign an Informed Consent Document or Assent, if applicable.
* Vision correctable to 20/30 Snellen (feet) or better in each eye at distance with pre-study contact lenses.
* Manifest cylinder (at screening) less than or equal to 0.75 diopters (D) in each eye.
* Successful wear of clear/handling tint, single-vision spherical, bi-weekly/ monthly replacement soft contact lenses in both eyes during the past 2 months for a minimum of 5 days per week and 8 hours per day.
* Requires spherical contact lenses within the available range of powers (i.e.,-1.50D to -5.00D in 0.25D steps).
* Interested in wearing contact lenses that change the appearance of the color of the eyes.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, disease or abnormality that contraindicates contact lens wear (within 7 days of enrollment, or current).
* History of herpetic keratitis.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated including any use of topical ocular medications that would require instillation during contact lens wear, except for rewetting drops.
* Corneal vascularization greater than 1 millimeter (mm) of penetration.
* Habitual lenses worn in an extended wear modality (routinely sleeping in lenses overnight for 1 night per week or more) over the last 3 months prior to enrollment.
* Previous corneal or refractive surgery or irregular cornea.
* Monovision and monocular (only 1 eye with functional vision) or fit with only 1 lens.
* Anisometropia ≥1.50D (study contact lens prescription).
* History of intolerance or hypersensitivity to any component of the test articles.
* Eye injury or ocular or intra-ocular surgery within the last 6 months (excluding placement of punctal plugs).
* Participation in any clinical study within 30 days of Visit 1.
* Other protocol-specified exclusion criteria may apply.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Brand Lead, GCRA, Vision Care, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 10 Study Centers located in the US.
Pre-assignment Details: Of the 151 enrolled, 1 subject was exited as a screen failure prior to randomization. This reporting group includes all randomized subjects (150).
Groups:
- AIR OPTIX COLORS: Contact lenses with color printing worn bilaterally in a daily wear modality 5 days/week, 8 hours/day for 30 days.
- FreshLook COLORBLENDS: Contact lenses with color printing worn bilaterally in a daily wear modality 5 days/week, 8 hours/day for 30 days with a 2-week replacement.
Period: Overall Study
Arm/Group | AIR OPTIX COLORS | FreshLook COLORBLENDS
Started | 74 | 76
Dispensed | 72 (Two subjects were randomized but never dispensed study lenses.) | 74 (Two subjects were randomized but never dispensed study lenses.)
Completed | 71 | 71
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Randomized in Error | 1 | 0
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects / eyes exposed to any test articles evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | AIR OPTIX COLORS | FreshLook COLORBLENDS | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (7.91) | 29.4 (7.62) | 29.7 (7.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 60 | 127
  Male | 5 | 14 | 19

OUTCOME MEASURES:

1. Primary Outcome: Lens Comfort Likert Response at Day 30
Description: Subject indicated agreement with the following statement, "These lenses provided the same excellent comfort at the end of the month as they did at the beginning of the month" using a 4-point Likert scale, where 1=Strongly disagree, 2=Disagree; 3=Agree; 4=Strongly agree. The Top 2 responses (agree, strongly agree) were calculated and reported as a percentage of all responses. Both eyes were rated together. This outcome measure was prespecified for the AIR OPTIX COLORS arm only.
Time Frame: Day 30
Population: This analysis population includes all randomized subjects excluding those who met the critical deviation criteria as specified in the Deviations and Evaluability Plan (DEP).
Measure: Number; unit: percentage of subjects
Arm/Group | AIR OPTIX COLORS
Number analyzed (Participants) | 70
percentage of subjects | 81.4

2. Secondary Outcome: Lens Comfort Likert Response at Day 14
Description: Subject indicated agreement with the following statement, "These lenses provided the same excellent comfort at the end of two weeks as they did at the beginning of the two weeks" using a 4-point Likert scale, where 1=Strongly disagree, 2=Disagree; 3=Agree; 4=Strongly agree. The Top 2 responses (agree, strongly agree) were calculated and reported as a percentage of all responses. Both eyes were rated together. This outcome measure is prespecified for the AIR OPTIX COLORS arm only.
Time Frame: Day 14
Population: This analysis population includes all randomized subjects with data at visit excluding those who met the critical deviation criteria as specified in the Deviations and Evaluability Plan (DEP).
Measure: Number; unit: percentage of subjects
Arm/Group | AIR OPTIX COLORS
Number analyzed (Participants) | 69
percentage of subjects | 89.9

3. Secondary Outcome: Lens Comfort 1-10 Scale Response
Description: Subject was instructed, "Please rate your comfort with the study lenses," using a scale from 1-10, where 1=poor and 10=excellent. Both eyes were rated together.
Time Frame: Day 30
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AIR OPTIX COLORS | FreshLook COLORBLENDS
Number analyzed (Participants) | 70 | 70
units on a scale | 8.0 (1.99) | 7.3 (2.19)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (3 months). AEs were reported by the subject and/or observed by the investigator as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the medical device.
Groups:
- Pre-treatment: Includes all subjects prior to the exposure to the investigational or control products
- AIR OPTIX COLORS: Includes all eyes exposed to AIR OPTIX® COLORS contact lenses
- FreshLook COLORBLENDS: Includes all eyes exposed to FreshLook® COLORBLENDS® contact lenses
Arm/Group | Pre-treatment | AIR OPTIX COLORS | FreshLook COLORBLENDS
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/144 | 0/148
Other Adverse Events (participants affected / at risk) | 0/151 | 0/144 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.